CLINICAL TRIAL: NCT06819202
Title: Effect of Hyperbaric Oxygen Therapy on Patients With Sudden Sensorineural Hearing Loss and Coagulation Function
Brief Title: Effect of Hyperbaric Oxygen Therapy(HBOT) on Patients With Sudden Sensorineural Hearing Loss(SSNHL) and Coagulation Function
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yuting (Other)
Responsible Party: Sponsor-Investigator, Sun Yuting, PhD student, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Other Study IDs: PTEC-A-2025-1(S)-1
Record Dates: First submitted 2025-01-25; First posted 2025-02-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sudden Sensorineural Hearing Loss (SSNHL); Hyperbaric Oxygen Therapy
MeSH Terms: conditions — Hearing Loss, Sudden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hyperbaric oxygen treatment — HBO therapy is the process of inhaling 100% pure oxygen in an environment above one atmosphere (pressure range: 2.0-3.0 absolute atmospheres) to treat a disease.

SUMMARY:
The objective of this observational study was to understand the effect of HBO on patients with SSNHL and its association with coagulation function and prognosis.

The main question it aims to answer is whether HBO therapy can improve outcomes and coagulation function in patients with SSNHL.

The prognosis of SSNHL patients receiving HBO and SSNHL patients not receiving HBO were compared

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for sudden deafness in the American Academy of Otolaryngology Head and Neck Surgery 2019 Clinical Practice Guidelines for Sudden Deafness;
* Aged 18-75 years old;
* Patients with unilateral sudden deafness for the first time, and the onset time is less than 2 weeks.

Exclusion Criteria:

* Patients with other ear diseases, such as auditory trauma, barotrauma, retrocochlear disease, bilateral hearing loss, history of chronic otitis media in the same ear, and history of surgery in the same ear;
* Patients with serious primary diseases such as heart, liver, kidney dysfunction and hematopoietic system diseases;
* Pregnant and nursing patients;
* Accompanied by serious mental illness;
* Patients with incomplete clinical data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2022 to September 2024, in Putuo Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Otolaryngology Hospital Affiliated to Fudan University, Xinhua Hospital affiliated to Shanghai Jiao Tong University or Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, treating patients with sudden sensorineural deafness.
Sampling Method: Probability Sample
Enrollment: 1309 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Hearing recovery rate | From onset to 3 months after treatment
  The rate of hearing recovery in patients with all levels of hearing loss at completion of treatment and at 3 months after termination of treatment was assessed according to the WHO Hearing Loss Rating Criteria 2021 to determine the success of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Traditional Chinese Medicine, Shanghai, Putuo, China

IPD SHARING:
Plan to Share IPD: No